CLINICAL TRIAL: NCT01162018
Title: Acupuncture for Sleep Disruption in Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, David Spiegel, Jack, Samuel and Lulu Willson Professor in Medicine, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BRSADJ0020; 1P30AT005886-01 (NIH); SU-04082010-5642 (Other: Stanford University)
Record Dates: First submitted 2010-07-02; First posted 2010-07-14 (Estimated); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Sleep Initiation and Maintenance Disorders; Breast Cancer
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Breast Neoplasms | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupuncture Arm (Experimental)
  Interventions: Procedure: acupuncture
- Sham Acupuncture (Sham Comparator): Sham Acupuncture
  Interventions: Other: placebo

INTERVENTIONS:
Procedure: acupuncture — The eligible women would be randomized and stratified by sleep problems to two arms: (Acupuncture Arm vs. Sham Acupuncture) with a goal of having 48 patients complete the study (we anticipate about 20% attrition rate). The study interventions will begin after patients completed their treatment. The placebo control for acupuncture will be a validated sham acupuncture control Assessments will be made with daily diaries and with weekly questionnaires. There are ten sessions each lasting approximately 20 minutes. All participants will have PSG data collected.
  Arms: Acupuncture Arm
Other: placebo
  Arms: Sham Acupuncture

SUMMARY:
The proposed study will recruit 60 women with breast cancer who finished undergoing treatment who complain of persistent insomnia problems that began with onset of their cancer diagnosis. The eligible women would be randomized and stratified by sleep problems to two arms: (Acupuncture Arm vs. Sham Acupuncture) with a goal of having 48 patients complete the study (we anticipate about 20% attrition rate). The study interventions will begin after patients completed their treatment. The placebo control for acupuncture will be a validated sham acupuncture control Assessments will be made with daily diaries and with weekly questionnaires. PSG data will be collected on the subsample of the population. Data will be gathered via pencil-and-paper measures before, during, immediately following, one month following the completion of treatment and six months after the conclusion of treatment. In addition, actigraphy data (objective sleep continuity data) will be acquired prior to and following treatment

ELIGIBILITY:
Inclusion Criteria:

* Females diagnosed with breast cancer who are not currently undergoing cancer treatment (hormonal treatment is permitted).
* The last cancer treatment ≥ 2 weeks prior to screening.
* ≥ 21 years of age.
* Able to understand written and spoken English.
* Have a habitual bedtime between 9:00 pm and 3:00 am and a habitual rise time between 4:00 am and 11 am.
* Meet DSM-IV criteria for insomnia (determined by the of the Duke Structured Interview of Sleep Disorders) with duration ≥ 1 month by Screening.
* Willingness to discontinue the use of any current sleep aides (prescription, OTC, or naturopathic agents).
* Properly executed Informed Consent.
* Karnofsky Performance Scale Index score ≥ to 70, (patients who score between 61-69 might be included per PI's evaluation).
* Insomnia Severity Index (ISI) > 8 at Screening.
* Able to travel to Stanford University and vicinity for assessments and acupuncture treatments.

Exclusion Criteria:

* Unstable medical or psychiatric illness (eMINI, current or within the last 5 years).
* Exposure to acupuncture within 6 months prior to screening.
* Currently pregnant or nursing.
* History of substance abuse or meet criteria for current alcohol abuse or dependence.
* Center for Epidemiological Studies Depression Scale (CES-D) >27 at Screening. Meet criteria for sleep apnea, restless legs syndrome or Circadian Rhythm Sleep Disorder on the basis of the Duke Structured Interview of Sleep Disorders (DSISD) or STOP-BANG is ≥ to 3.
* Major surgery within 4 weeks prior to first acupuncture treatment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 65 (Actual)
Dates: Start 2011-02; Primary Completion 2012-07 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Fatigue reduction | 1 month and 3 months post final acupuncture treatment
Quality of life in breast cancer survivors after acupuncture | 1 month and 6 months post final acupuncture treatment
  Quality of life in breast cancer survivors after acupuncture will be measured through questionnaire using 28 item scale of functional assessment of chronic illness therapy- fatigue subscale (FACIT-F) version 4. Total score ranges from 0 to 108. A higher score indicates better quality of life.
Insomnia reduction | 1 month and 3 months post final acupuncture treatment

CONTACTS AND LOCATIONS:
Overall Officials: David Spiegel, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States